CLINICAL TRIAL: NCT07184970
Title: Prostate Recurrence Detection Using Imaging With PSMA PET/MRI Post-high Intensity Focused Ultrasound
Brief Title: PRISM Study: Prostate Recurrence Detection Using Imaging With PSMA PET/MRI Post-high Intensity Focused Ultrasound
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 24-01935
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men with Prostate Cancer: Patients undergoing High-Intensity Focused Ultrasound (HIFU) for focal therapy of prostate cancer. Participants will be followed for one-year post-treatment, with regular monitoring through various clinical assessments.

SUMMARY:
The purpose of this study is to compare the sensitivity of PSMA PET/MRI and standard MRI in detecting focal therapy failure in the prostate one year after High-Intensity Focused Ultrasound (HIFU) treatment. Specifically, the study aims to evaluate whether PSMA PET/MRI offers a higher sensitivity than MRI alone for identifying recurrence or failure in patients undergoing focal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male patients 40-95 years of age with biopsy-confirmed localized prostate cancer.
* Grade Group ≥2 (Gleason score 3+4 or higher).
* Unifocal disease visible on mpMRI.
* Patients undergoing HIFU as part of their standard of care
* PSA <20 ng/mL.
* No metastatic disease on PSMA PET/CT
* Willingness to comply with follow-up protocols (PSA testing, imaging, biopsies).

Exclusion Criteria:

* Evidence of metastatic disease on PSMA PET/CT.
* Allergy to POSLUMA or gadolinium.
* Inability to tolerate MRI due to claustrophobia or posture/back-hip issues.

Ages: 40 Years to 95 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Only male patients will be included in this study. The expected age range will be 40-95. There is no enrollment restrictions based upon race or ethnic origin.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of PSMA PET/MRI | Month 12
  Sensitivity of PSMA PET/MRI for detecting clinically significant prostate cancer at 12 months post HIFU, defined as the portion of patients with clinically significant cancer on the 12-month biopsy (reference standard) who had a positive PSMA PET/MRI.
Oncologic Control | Month 12
  Oncologic control at 12 months, defined as the absence of cancer, determined by the scheduled biopsy at 12 months.

SECONDARY OUTCOMES:
Portion of patients achieving a PSA reduction greater than 50% | Month 3, Month 6, Month 12
  The portion of patients achieving a PSA reduction greater than 50% from pre-HIFU baseline measured at 3 months, 6 months, and every 6 months post-HIFU.
Change in IPSS (International Prostate Symptom Score) | Baseline, Month 12
  The IPSS (International Prostate Symptom Score) assesses lower urinary tract symptoms (LUTS). A total IPSS score of 1-7 is considered mild, 8-19 moderate, and 20-35 severe.
Change in SHIM (Sexual Health Inventory for Men) Score | Baseline, Month 12
  The SHIM (Sexual Health Inventory for Men) score measures erectile dysfunction (ED). A SHIM score of 22-25 indicates no ED, 17-21 is mild, 12-16 mild to moderate, 8-11 moderate, and 1-7 severe ED.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Phin Tan, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: weiphin.tan@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to weiphin.tan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.